CLINICAL TRIAL: NCT06086808
Title: Effect Of Resistance Training On Physical Fitness, Cognitive Ability, And Academic Performance In Young Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/01612 Tahreem Nisar
Record Dates: First submitted 2023-10-04; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Young Adults
Keywords: Academic Performance; Cognitive Function; Exercise Training; Physical Fitness; Resistance Training
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Concurrent Parallel Randomized Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Resistance Training Group
  Interventions: Other: Resistance Training
- Group B (Active Comparator): General Fitness and Toning Group
  Interventions: Other: General Fitness and Toning

INTERVENTIONS:
Other: Resistance Training — A resistance training program will be used as a progressive, high-intensity protocol. The training stimulus will be provided using free weights. The exercises will consist of bench presses, biceps curls, triceps extensions, Latissimus Dorsi pull-down exercises, hamstring curls, and calf raises. The intensity of the training stimulus will be at a working range of 6 to 8 repetitions (2 sets). The training stimulus will subsequently be increased using the 7-RM (repetition maximum) method when 2 sets of 6 to 8 repetitions are completed with proper form and without discomfort. Other key strength exercises will include mini-squats, mini-lunges, and lunge walks. The number of sets completed and the load lifted for each exercise will be recorded for each participant in every class.
  Arms: Group A
Other: General Fitness and Toning — The general fitness and toning program will consist of stretching exercises, range-of-motion exercises, basic core-strengthening exercises, balance exercises, and relaxation techniques. Key balance exercises will include tandem stand, tandem walking, and single leg stance (eyes opened and closed). No additional loading (e.g., hand weights or resistance bands) will be applied to any of the exercises. This group will serve to control for confounding variables such as physical training received by traveling to the training centers, social interaction, and changes in life style secondary to study participation.
  Arms: Group B

SUMMARY:
The goal of this study is to determine the effect of resistance training on physical fitness, cognitive ability, and academic performance in young adults. This would be a randomized controlled trail in which participants will be randomly allocated in to two groups. One group will perform resistance training and other group will perform balance and general body toning exercises.

DETAILED DESCRIPTION:
In recent years, the relationship between physical fitness, cognitive ability, and academic performance has garnered significant attention in the fields of education, psychology, and sports science. Young adulthood represents a critical developmental period characterized by substantial physical, cognitive, and psychological changes. During this phase, individuals are often engaged in academic pursuits, which makes understanding the impact of various interventions on physical fitness, cognitive ability, and academic performance especially relevant.

While individual studies have explored the effects of resistance training on physical fitness, cognitive ability, and academic performance separately, there remains a gap in the literature concerning a comprehensive understanding of their interconnectedness in the context of young adults. This study aims to bridge this gap by investigating the potential causal relationship between resistance training and these multifaceted outcomes.

This randomized controlled trial will recruit participants from young population. Study participants will be randomized into two groups: Group-A and Group-B. Group-A participants would receive resistance training for 3 consecutive months, while Group-B participants would follow general fitness and body toning exercises. Physical fitness, cognitive ability and academic performance will be measured at the baseline and after the termination of intervention program.

ELIGIBILITY:
Inclusion Criteria:

* School going children between the ages of 12 to 17 year

Exclusion Criteria:

* Participants with any recent musculoskeletal injury that hasn't healed.
* Any deformity or disability that could affect the participant's ability to perform physical activity.
* Any systemic disease/disorder that could affect the physical and cognitive performance of the participants.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Isometric Strength (lbs) | Baseline and after end of the intervention (3 months)
  Isometric Strength will be assessed using a Hand-held Dynamometer measuring isometric contraction force in pounds (lbs).
Endurance | Baseline and after end of the intervention (3 months)
  Endurance will be assessed using the Yo Yo Intermittent Recovery Level 1 Test ranging from speed level 5 (lightest) to speed level 23 (hardest).
Agility | Baseline and after end of the intervention (3 months)
  Agility will be assessed using Illinois Agility Run Test (Time to complete it in seconds).
Balance | Baseline and after end of the intervention (3 months)
  Balance will be assessed using Star Excursion Balance Test (distance in each direction).
Stroop Test | Baseline and after end of the intervention (3 months)
  Stroop test will be used to assess cognitive function (number of items completed during each task).
Trail Making Test | Baseline and after end of the intervention (3 months)
  Trail Making Test will be used to assess cognitive function (time spent to complete the task).
Verbal Digit Span Test | Baseline and after end of the intervention (3 months)
  Verbal Digit Span Test will be used to assess cognitive function (number of digits recalled correctly).
Academic Performance | Baseline and after end of the intervention (3 months)
  Academic performance will be assessed using previous and subsequent school grades of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Noman Sadiq, MS-SPT, Principal Investigator — Riphah International University, Islamabad.
Locations (1):
- Riphah International University (RIU), Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No